CLINICAL TRIAL: NCT06267339
Title: Effects of Transcranial Random Noise Stimulation on Motor Learning in Typically Developing Adolescents
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Burke Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TD_tRNS
Record Dates: First submitted 2024-01-30; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Children
Keywords: typically developing children; motor learning; controls; grasp; reach
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Grasp Task (Experimental): Participants will practice a fine motor grasping task for 20 min during tRNS or sham stimulation.
  Interventions: Device: transcranial random noise stimulation; Device: Sham stimulation
- Reach Task (Experimental): Participants will practice a reaching task for 20 min during tRNS or sham stimulation.
  Interventions: Device: transcranial random noise stimulation; Device: Sham stimulation

INTERVENTIONS:
Device: transcranial random noise stimulation — This intervention will give children tRNS during reaching or grasping repetitive movements.
Device: Sham stimulation — This intervention will give children sham stimulation during reaching or grasping repetitive movements.

SUMMARY:
The goal of this study is to compare motor learning rates on two different tasks, when combined with non-invasive brain stimulation.

DETAILED DESCRIPTION:
We will apply transcranial random noise stimulation or sham stimulation. During tRNS, participants will complete a grasping task or a reaching task. Each participant will complete both tasks, with a wait period between each task. Task order will be randomized, such that half the group will begin with each task. We will compare task scored before vs. after tRNS, for each task. This will be a measure of motor learning.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-17 years
* Ability to follow two-step instructions
* Provides informed consent

Exclusion Criteria:

* Presence of illness, disease

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Grasp score | Immediately before vs. Immediately after brain stimulation
  Participants will be asked to perform a grasping task, scored by number of pegs placed in a board.
Change in Reach score | Immediately before vs. Immediately after brain stimulation
  Participants will be asked to perform a reaching task to stack cups, scored by time taken to stack all cups.

SECONDARY OUTCOMES:
Change in Graded Redefined Assessment of Strength, Prehension assessment (GRASSP) | Immediately before vs. Immediately after brain stimulation
  Participants will be asked to perform the GRASSP, scored by tallying points according to the test parametrics.
Change in score on second reaching task | Immediately before vs. Immediately after brain stimulation
  Participants will be asked to perform a reaching task to stack cups in a different pattern from Primary Outcome #2, scored by time taken to stack all cups.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Friel, PhD, Principal Investigator — Burke Neurological Institute
Locations (1):
- Burke Neurological Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We will upload de-identified data onto our website and the NIH data sharing website (DASH).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be uploaded within 2 months of study completion and will be available in perpetuity.
Access Criteria: Potential users will need to join DASH to access our data. Anyone who completes the DASH registration will be able to access our data.
URL: https://dash.nichd.nih.gov/